CLINICAL TRIAL: NCT00378131
Title: A 12-Week, Double-Blind, Randomized, Placebo-Controlled, Parallel Group Phase II Study Comparing the Safety, Tolerability and Beneficial Effects of Daily Doses of RC-1291 and Placebo in Patients With Cancer Anorexia/Cachexia
Brief Title: Placebo Controlled, Randomized Safety and Efficacy Study of RC-1291 in Cancer Anorexia/Cachexia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helsinn Therapeutics (U.S.), Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC-1291-206
Record Dates: First submitted 2006-09-18; First posted 2006-09-19 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Cancer Cachexia
MeSH Terms: interventions — RC-1291

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: placebo
- 2 (Experimental): RC-1291 50mg
  Interventions: Drug: RC-1291
- 3 (Experimental): RC-1291 100mg
  Interventions: Drug: RC-1291

INTERVENTIONS:
Drug: RC-1291
  Arms: 2; 3
Drug: placebo
  Arms: 1

SUMMARY:
Activation of Ghrelin receptors have been demonstrated to stimulate appetite. RC-1291 HCl, by virtue of its ghrelin like activity and Growth Hormone releasing effects may have a dual role in the reversal of cancer induced anorexia and cachexia. This placebo controlled study will evaluate the safety and efficacy of RC-1291 HCl in cancer patients with cachexia.

DETAILED DESCRIPTION:
Anorexia and cachexia are devastating complications in late-stage cancer patients and is strongly associated with mortality in these patients. Activation of Ghrelin receptors have been demonstrated to stimulate appetite. RC-1291 HCl, by virtue of its ghrelin like activity and Growth Hormone releasing effects may have a dual role in the reversal of cancer induced anorexia and cachexia. This placebo controlled study will evaluate the safety and efficacy of RC-1291 HCl in cancer patients with anorexia and cachexia.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling patients greater than 18 years of age with incurable, histologically diagnosed cancer.
* Involuntary loss of body weight greater than 5% within the past 6 months

Exclusion Criteria:

* Presently hospitalized or in a nursing care facility.
* Inability to increase food intake from secondary causes.
* Liver disease
* If female-pregnant, breast-feeding or of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-09; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Body weight; Lean body mass; Functional performance | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: William Polvino, MD, Study Director — Helsinn Therapeutics (U.S.), Inc
Locations (17):
- United States (17):
  - Palo Verde Hematology Oncology, Ltd., Glendale, Arizona
  - San Diego Pacific Oncology & Hematology Associates, Encinitas, California
  - Sant P. Chawla, MD, Santa Monica, California
  - Melbourne Internal Medicine Associates, Melbourne, Florida
  - Southwest Oncology Associates, Lafayette, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - Chesapeake Oncology Hematology Associates, PA, Glen Burnie, Maryland
  - Beth Israel Cancer Center, New York, New York
  - Charleston Cancer Center, Charleston, South Carolina
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - South Carolina Cancer Specialists, Hilton Head Island, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Cancer Outreach Associates, Abingdon, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Multicare Health System, Tacoma, Washington
  - Northwest Medical Specialties, Tacoma, Washington